CLINICAL TRIAL: NCT05888584
Title: Improving Access and Recruitment to Clinical Trials for Lung Cancer Patients
Acronym: LungI-ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: De Montfort University (Other)
Responsible Party: Principal Investigator, Dr Cathy Henshall, Professor Catherine Henshall, Oxford Brookes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRAS project ID: 325757
Record Dates: First submitted 2023-05-12; First posted 2023-06-05 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer
Keywords: lung cancer; nurses; research; clinical trials; recruitment; access
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention tool (Experimental): A research recruitment tool will be available in paper and online formats and will include information on finding out about LC clinical trials, the role of research teams, embedding research into multidisciplinary team meetings and health needs assessments, communication pathways, signposting LCPs, practical considerations and reaching underrepresented groups. The tool will be used by lung cancer nurses in their daily practice as an aid to support their discussions with lung cancer patients about clinical trial opportunities. They will be asked to complete a survey at three time-points (baseline, three and six months) to measure their self-efficacy, knowledge, confidence and awareness in talking to lung cancer patients about clinical trials.
  Interventions: Other: Research readiness tool
- Control (No Intervention): Lung cancer nurses will undertake usual care. They will be asked to complete a survey at three time-points (baseline, three and six months) to measure their self-efficacy, knowledge, confidence and awareness in talking to lung cancer patients about clinical trials.

INTERVENTIONS:
Other: Research readiness tool — Online/paper based tool for use by nurses to aid discussions with lung cancer patients about clinical trials opportunities.
  Arms: Intervention tool

SUMMARY:
There are ~85,000 lung cancer patients (LCPs) in the UK; yet only around 8% were recruited into clinical trials in 2021/22. LCPs need opportunities to take part in clinical trials to access new treatments, increasing their quality of life, treatment choices and life expectancy.

Discussions with nurses can help patients make better treatment decisions, improving experiences of care. However, research has shown that lung cancer nurses (LCNs) often feel unable to discuss participation in trials with patients due to lack of knowledge, confidence, time and training.

This study aims to develop and test a research recruitment tool for LCNs, to support LCPs to enter clinical trials.

Objectives include to:

* Explore reasons for low uptake of LCPs into clinical trials
* Develop a tool for LCNs to talk to patients about clinical trials
* Test whether the tool improves the number and quality of discussions nurses have with LCPs about clinical trials

The study has four phases:

Phase 1: A literature review will identify problems that make clinical trial uptake difficult for LCPs, carers and clinicians

Phase 2: Six group discussions with LCNs, patients and carers will explore issues that create potential barriers for patients taking part in clinical trials. The groups will take place online, last approximately one hour and be recorded.

Phase 3: Part 1&2 findings will help us develop a LCN research recruitment tool. The tool will contain information on how nurses obtain information about LC clinical trials, research teams, communication issues, practical issues and how to reach LCPs.

Phase 4: The research recruitment tool will be tested in four UK NHS hospitals. A survey will identify any changes in nurses' clinical trials awareness and confidence before and after using the tool. Interviews with LCNs, patients and carers will explore their views on the tool, clinical trials participation and experiences of care.

DETAILED DESCRIPTION:
Background: Patients who discuss taking part in research and those that go on to participate have better outcomes and experiences. Reported trial benefits for patients include greater access to new drugs; disease control; improved survival; enhanced quality of life; more intensive follow up and monitoring; better symptom management; enhanced care and support; and patient empowerment. In cancer care, the rate at which targeted treatments are translated into clinical practice for use by LCPs is reliant on accessible clinical trial opportunities; however, trial uptake remains low. Recruitment to research within the UK National Health Service (NHS) is challenging and COVID-19 saw a 59% reduction in cancer patients entering clinical trials in England, from 67,057 in 2017/18 to 27,734 in 2020/2021 [7,8]. Resultingly, the Institute of Cancer have recommended that trial information is made accessible and understandable to patients and that clinical staff have conversations about trials early in the treatment pathway.

Being assigned a LC clinical nurse specialist is associated with better experiences of care and studies have found that discussions nurses have with patients about clinical trial enrolment play a key role in decision-making and recruitment. However, LCNs often feel unable to discuss clinical trials with patients due to a lack of knowledge and confidence, time, expertise and training. Key barriers to trial recruitment include screening complexities; lack of resources, staff, skills and equipment; time; limited clinician awareness; perceived administrative burdens, concerns over trial suitability; inadequate information communicated to patients and clinicians and complex trial terminology. It is recommended that clinical trials are more closely integrated into clinical practice and that staff are adequately trained to support clinical research.

Study design: This mixed methods study consists of the following phases:

Phase 1: A systematic review of the best scientific literature will identify challenges and barriers to clinical trial recruitment amongst LCPs, carers and clinicians. PRISMA reporting guidelines will be followed.

Phase 2: Six qualitative focus groups with lung cancer patients, carers, lung cancer nurses and other members of the multidisciplinary team (MDT) will explore challenges and facilitators to LCPs' clinical trial entry. Focus group participants will be recruited through the participating sites lung cancer nursing teams.

Eligible clinician participants (nurses and other MDT staff) will be contacted through lead LCNs at participating sites (see phase 4), who will share invitation letters and participant information leaflets with their teams. If they are happy to proceed a researcher will organise a time, date and place with participants to proceed with the focus group. Participants will also be recruited through LCNUK and the National Institute for Health Research (NIHR) Local Clinical Research Networks.

Patients and carers will be recruited through the NCRI consumer forum and other cancer patient/carer networks, including RCLCF and Mesothelioma UK. LCNs at participating NHS sites will also share invitation letters and information leaflets with LCPs, inviting them to take part. If they are happy to proceed the researcher will organise a time, date and place with participants to proceed with the focus group. The study will also be promoted via social media channels such as Twitter, Healthcare Unlocked and closed Facebook groups. We intend to recruit ~48 participants to focus groups (eight per group); three focus groups will be with LCNs, research nurses and multidisciplinary team members from district general hospitals (DGHs) and tertiary centres, and two with LCPs and carers. A final group will include clinicians from the Christie and Royal Marsden cancer centres, where recruitment to trials is higher than in DGHs and tertiary centres, to identify transferable elements of best practice. Focus groups will be held remotely, via the online Zoom platform.

Focus groups facilitated by two researchers, will last one hour, and will be recorded and transcribed. Data will be thematically analysed using the Framework Method, to enable comparisons across groups to be identified and themes generated.

Phase 3: Phase 1&2 findings will inform development of the LCN research recruitment tool. The tool, available in paper and online formats, will include information on finding out about LC clinical trials, the role of research teams, embedding research into multidisciplinary team meetings and health needs assessments, communication pathways, signposting LCPs, practical considerations and reaching underrepresented groups. Tool development will be guided by the Trial Steering Group (TSG), with representation from LC patient and public involvement (PPI) members, LCNs, multidisciplinary research and clinical teams. The tool will be tested for face and content validity by ~10 LCNs who participated in Phase 2, and ~4 PPI representatives. Relevant feedback will be used to make modifications to the tool.

Phase 4 pilot: Participants in the pilot study will pilot the research recruitment tool for proof of concept across four UK NHS sites, including tertiary centres and DGHs: Oxford, Derby&Burton, Lanarkshire, Nottinghamshire. An additional two NHS sites, Surrey and Birmingham, will act as controls.

Each site's LCNs (n=36) will be invited to participate through their senior nurse manager who will provide eligible nurses with an online invitation letter and participant information sheet (PIS). If they are happy to proceed the researcher will organise a time, date and place with participants for the pilot phase of the study. Nurse participants will then have a briefing session, where the pilot study purpose will be explained. LCNs at the pilot sites (n=24) will be provided with a training session on using the tool, before implementing it in their teams for six months.

Survey data will be collected from each LCN (n=36) at baseline, three and six months and LCN's will reconsent electronically, via the Qualtrics survey platform, prior to completing each online survey. The survey will collect information on the following: 1) Items from the validated General Perceived Self-Efficacy Scale will measure LCNs' self-efficacy (primary outcome measure) in relation to their research roles 2) The number of LCPs each LCN has approached to discuss clinical trial opportunities will be recorded 3) Likert style survey data on LCNs' knowledge, confidence and awareness of clinical trials will be collected. These questions will be developed from phase 1&2 findings and tested for reliability and validity by TSG members. The repeated tests measure ANOVA will compare survey responses between baseline, three and six months. Between groups ANOVA will compare differences in scores between pilot and control sites. No formal sample size calculation is required as this is a pilot study; however, all LCNs across the six sites will be invited to take part (n~36).

Towards the end of the pilot, eight LCNs who have been taken part in the pilot will be invited, via an invitation letter and participant information sheet provided by the research team, to attend a 30-minute interview, via the online Zoom platform, or via telephone, to explore the tool's acceptability, in terms of ease of use and impact on recruitment.

Eight patients/carers who have joined clinical trials at the pilot sites will also be interviewed remotely, via the online Zoom platform or by telephone to explore their clinical trial experience and its impact on quality of life, care satisfaction, self-efficacy and symptom control will be explored. This will provide valuable information on the tool's impact on LCP experience.

ELIGIBILITY:
Healthcare staff Phase 2:

Inclusion Criteria:

* Actively involved in the clinical care pathways of lung cancer patients
* Working at one of the six participating NHS trusts
* Age between 18-65 years of age

Exclusion criteria:

* Not actively involved in frontline clinical care
* Not involved in caring for lung cancer patients for at least 30% of their

Patients/carers:

Inclusion criteria:

* Must have a current diagnosis of lung cancer (any stage) or be the named carer of a person with a lung cancer diagnosis
* Under the care of (or caring for) one of the participating NHS Trusts lung cancer teams
* Aged 18 or over

Exclusion criteria:

* Mesothelioma diagnosis or caring for someone with a mesothelioma diagnosis
* Unable to provide informed consent

Phase 4 Healthcare professionals

Inclusion criteria:

* Registered nurse with Nursing and Midwifery Council
* Actively involved in the clinical care pathways of lung cancer patients
* Working at one of the six participating NHS trusts
* Age between 18-65 years of age

Exclusion criteria:

* Not actively involved in frontline clinical care
* Not involved in caring for lung cancer patients for at least 30% of their role
* Employed as a lung cancer research delivery nurse

Patients/carers:

Inclusion criteria:

* Current diagnosis of lung cancer (any stage) or be the named carer of a person with a lung cancer diagnosis
* Aged 18 or over
* Consented to (or carer of someone who has consented to) a clinical trial since start of pilot study
* Receiving care (or carer for someone receiving care) in one of the four NHS sites piloting the research readiness tool

Exclusion criteria:

* Mesothelioma diagnosis or caring for someone with a mesothelioma diagnosis
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
self-efficacy | six months
  Data will be collected from each lung cancer nurse (n=36) at baseline, three and six months. Items from the validated General Perceived Self-Efficacy Scale (GSE) will measure LCNs' self-efficacy in relation to their research.
  The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.

SECONDARY OUTCOMES:
research contacts with lung cancer patients | six months
  Data will be collected from each LCN (n=36) at baseline, three and six months on the number of lung cancer patients each lung cancer nurse has approached to discuss clinical trial opportunities
lung cancer nurses' clinical trials knowledge | six months
  Data will be collected from each lung cancer nurse (n=36) at baseline, three and six months on their knowledge of clinical trials. Data will be collected via a non-validated Likert style survey with five options ranging from 'strongly agree' to 'strongly disagree'.
lung cancer nurses' clinical trials confidence | six months
  Data will be collected from each lung cancer nurse (n=36) at baseline, three and six months on their confidence in talking to lung cancer patients about clinical trials. Data will be collected via a non-validated Likert style survey with five options ranging from 'strongly agree' to 'strongly disagree'.
lung cancer nurses' clinical trials awareness | six months
  Data will be collected from each lung cancer nurse (n=36) at baseline, three and six months on their awareness of lung cancer clinical trials opportunities. Data will be collected via a non-validated Likert style survey with five options ranging from 'strongly agree' to 'strongly disagree'.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Henshall, PhD, Principal Investigator — Oxford Brookes University
Locations (9):
- United Kingdom (9):
  - Derby and Burton NHS, Derby, Derbyshire
  - St Bartholomews Hospital NHS, London, Greater London
  - The Royal Marsden NHS, London, Greater London
  - The Christie NHS, Manchester, Greater Manchester
  - Sherwood Forest NHS, Nottingham, Nottinghamshire
  - Oxford University Hospitals, Oxford, Oxfordshire
  - Royal Surrey County Hospital, Guildford, Surrey
  - Sheffield Teaching Hospitals NHS, Sheffield, Yorkshire
  - Lanarkshire NHS, Glasgow

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with researchers outside of the study team.